CLINICAL TRIAL: NCT00941876
Title: An Evaluation of Integration of Family Planning Into HIV/AIDS Care and Treatment Clinics in Tanzania
Brief Title: Integration of Family Planning and HIV Services in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Mackenzie Green, FHI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10121
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infection; HIV Infections
Keywords: AE; adverse event; AIDS; acquired immunodeficiency syndrome; ALT (SGPT); alanine aminotransferase; ART; antiretroviral therapy; AST (SGOT); aspartate aminotransferase; DCF; data collection forms; DMC; Data Monitoring Committee; FDA; (U.S.) Food and Drug Administration; GCP; Good Clinical Practice guidelines; HB sAg; Hepatitis B surface antigen; ICH; International Conference of Harmonisation; IND; Investigational New Drug Application; IRB; Institutional Review Board; IU; International units; mg; milligram(s); mm3; cubic millimeter(s); PCR; polymerase chain reaction; SAE; serious adverse event; µg; microgram; ULN; upper limit of the normal range; WB; Western Blot; To inform the Ministry of Health strategy for integrating FP and HIV/AIDS Care and Treatment Services in Tanzania; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A. Facilitated Referral (Experimental): Seven key steps carried out by CTC and FP staff to encourage completion of FP referral by CTC.
  Interventions: Behavioral: Facilitated Referral

INTERVENTIONS:
Behavioral: Facilitated Referral — Seven key steps carried out by CTC and FP staff to encourage completion of FP referral by CTC.

SUMMARY:
HIV positive women and couples have broad reproductive health needs that are not always met within HIV services. The integration of family planning (FP) services into Tanzania's HIV Care and Treatment Clinics (CTC) will address the fertility desires of CTC clients and ultimately result in the reduction of unintended pregnancies and HIV incidence. One strategy for integrating FP and CTC services is to use a "facilitated referral" model. Facilitated referrals are enhanced referrals for additional services that have been used in other settings and which are the preferred intervention strategy the Government of Tanzania would like to pilot test. This study will evaluate the feasibility, effectiveness, and costs of implementing a "facilitated referrals" intervention by examining FP use among female clients attending HIV/AIDS Care and Treatment Centers. This study will measure whether there is a reduction in unmet need for contraception among female CTC clients after the facilitated referral integration intervention has been implemented.

ELIGIBILITY:
Inclusion Criteria:

1. Female clients of Care & Treatment Clinics with CD4 counts >100, and are WHO Stage I - III. (CTC Clients)
2. Care and Treatment providers who provide services to clients (CTC Providers)
3. Care and Treatment supervisors who are the immediate in-charge supervisor for the CTC clinic. (CTC supervisor)
4. Family Planning providers who provide services to clients. (FP providers)
5. Family Planning supervisors who are the immediate in-charge supervisor for the FP clinic. (FP supervisor)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 864 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Proportion of female CTC clients with unmet need for contraception | Before intervention begins (baseline) and 3 months after full implementation of intervention

SECONDARY OUTCOMES:
Proportion of female CTC clients screened on fertility intentions and unmet need for contraception | Three months after full implementation of intervention
Proportion of female CTC clients provided counseling on contraception or safe pregnancy | Three months after full implementation of intervention
Proportion of female CTC clients who received referral slip for FP services | Three months after full implementation of intervention
Proportion of female CTC clients whose contraceptive use/fertility intentions are recorded on their patient record form | Three months after full implementation of intervention
Proportion of female CTC clients who are accompanied to FP services | Three months after full implementation of intervention
Proportion of female CTC clients who receive a FP method same-day or make an appointment for sterilization | Three months after full implementation of intervention
Proportion of referrals to FP services that are tracked by the FP clinic | Three months after full implementation of intervention
Incremental cost per clinic of adding facilitated referral process for FP to existing CTC services | First month of implementation
Descriptive data on the experiences and perception of CTC and FP providers and supervisors on how the facilitated referral for FP was feasible and effective within CTC services | Three months after full implementation of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joy N Bumgartner, MSW, PhD, Principal Investigator — FHI 360; Thecla W Kohi, PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Muhimbili University of Health and Allied Services, Dar es Salaam, Tanzania